CLINICAL TRIAL: NCT06614348
Title: A Randomized Controlled Study of Prednisolone Acetate Eye Drops for Pain Intervention in Second Eye Cataract Surgery
Brief Title: Prednisolone Acetate Eye Drops for Pain Intervention in Second Eye Cataract Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Huiyi Jin, Principal Investigator, Associate Chief Physician,, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCTR-2023C03
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Age Related Cataract; Pain Management During Cataract Surgery
Keywords: cataract surgery; pain; second-eye cataract surgery
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisolone acetate eye drop group (Experimental)
  Interventions: Drug: Prednisolone acetate eye drop group
- hyaluronic acid eye drop group (Placebo Comparator)
  Interventions: Drug: Sodium hyaluronate eye drops

INTERVENTIONS:
Drug: Prednisolone acetate eye drop group — Patients receive prednisolone acetate eye drops 4 times per 30min within 2 hours before cataract surgery
  Arms: Prednisolone acetate eye drop group
Drug: Sodium hyaluronate eye drops — Patients receive sodium hyaluronate eye drops 4 times per 30min within 2 hours before cataract surgery
  Arms: hyaluronic acid eye drop group

SUMMARY:
This study aims to evaluate the efficacy, safety, and potential mechanisms of prednisolone acetate eye drops for pain management in patients undergoing second-eye surgery for age-related cataracts.

Researchers will compare prednisolone acetate eye drops to sodium hyaluronate eye drops to see if prednisolone acetate eye drops work to relieve intraoperative and postoperative pain during second-eye cataract surgery.

Participants will:

1. Receive prednisolone acetate eye drops or sodium hyaluronate eye drop four drops within 2 hours before cataract surgery
2. Finish cataract surgery and routine postoperative follow-up
3. Pain questionnaire completed after cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* Age between 50-80 years old;
* A clear diagnosis of age-related cataract, having completed the first eye cataract surgery at our hospital, and planning to have the second eye cataract surgery with the same doctor;
* The interval between the two surgeries is ≤30 days;
* Capable of cooperating to complete iris optical coherence tomography angiography examination;
* Based on our team's previous research, a predictive scoring formula for pain during the second eye surgery has been derived (Predicted score = 1.36 + 4.93 * preoperative iris vessel area density - 0.24 * surgical interval (weeks)), and the calculated predicted score is >2.

Exclusion Criteria:

* History of ocular trauma, ocular surgery, uveitis, fundus disease, glaucoma, or recent history of episcleritis, keratitis, severe dry eye, and other ocular surface disease episodes;
* Participation in intraocular or systemic medication clinical trials within the past 6 months;
* Having an autoimmune disease or currently undergoing immunosuppressive therapy;
* Having a psychiatric disorder such as anxiety or depression;
* History of using glucocorticoid eye drops for treatment in the second eye within the past month;
* Long-term use of drugs that can cause intraoperative floppy iris syndrome, such as alpha-blockers;
* Severe complications occurred during or after the first eye surgery (e.g., posterior capsule rupture, zonular exercise, nuclear drop into the vitreous cavity, postoperative endophthalmitis, glaucoma, etc.).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10-08 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain scores measured by Visual Analogue Scale | Within one hour after surgery
  Within one hour after surgery, the investigator uses the Visual Analogue Scale (VAS) to allow the patient to self-assess the degree of pain. A movable ruler about 10 cm long is used, with one side unmarked and the other side marked with scales, with the ends labeled "0" for no pain and "10" for the most severe pain that is unbearable. The investigator holds the marked side of the ruler away from the patient, allowing the patient to mark the position on the ruler that represents their level of pain. The investigator then records the corresponding score based on the position marked by the patient.

SECONDARY OUTCOMES:
Comparison of pain during the second eye surgery to the first eye surgery | Within one hour after surgery
  Within one hour after the surgery, the investigator asks the patient to compare the pain experienced during the second eye surgery with that of the first eye surgery. The patient is asked to choose the most appropriate statement from the following: 1. I think the pain during the second eye surgery was worse than the first eye surgery; 2. I think the pain during the second eye surgery was less than the first eye surgery; 3. I think the pain during the second eye surgery was about the same as the first eye surgery; 4. I do not remember the pain during the first eye surgery; and the result is recorded by the investigator.
Expression levels of monocyte chemotactic protein-1 in the aqueous humor of surgical eyes | Within three months after surgery
  The aqueous humor is detected using a cytokine array according to the instructions of manufacturer.
Best Corrected Visual Acuity (BCVA) of the surgical eye | One month after surgery
  When testing Best Corrected Visual Acuity (BCVA) with the Snellen chart, first ensure that the patient is wearing the appropriate corrective lenses. Then ask the patient to stand 20 feet (6 meters) away from the chart. Instruct the patient to cover one eye with a hand, and test the uncovered eye. Starting from the top, have the patient read the smallest line of text they can see clearly. Record the vision of the smallest line that the patient can read completely and correctly.
Adverse events and severe adverse events | From enrollment to one month after surgery
  Adverse Events (AEs):
  Intraoperative complications: such as posterior capsule rupture, zonular dialysis, inability to implant an intraocular lens, etc.
  Postoperative infection: Infection at the surgical site, which may require additional antibiotic treatment or surgical intervention.
  Changes in vision: Decreased vision after surgery can occur even without apparent complications.
  Elevated intraocular pressure: Intraocular pressure may be temporarily or persistently elevated after surgery, necessitating medication or surgical intervention.
  Serious Adverse Events (SAEs):
  Retinal detachment, endopthalmitis, persistent high intraocular pressure, severe bleeding, dislocation of the lens or intraocular lens, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Huiyi Jin, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang Y, Du Y, Jiang Y, Zhu X, Lu Y. Effects of Pranoprofen on Aqueous Humor Monocyte Chemoattractant Protein-1 Level and Pain Relief During Second-Eye Cataract Surgery. Front Pharmacol. 2018 Jul 17;9:783. doi: 10.3389/fphar.2018.00783. eCollection 2018. PMID 30065652
- [Background] Cui L, Ma Y, Wang Y, Luo Q, Ding Q, Ge L, Lu S, Miao Y, Sun Q, Zou H, Jin H. Combination of iris vessel area density and surgery interval as the predictor of perceived pain during consecutive second-eye cataract surgery. J Cataract Refract Surg. 2023 Aug 1;49(8):858-863. doi: 10.1097/j.jcrs.0000000000001229. PMID 37350758